CLINICAL TRIAL: NCT03660774
Title: Evolving Treatment of Hemophilia's Impact on Neurodevelopment, Intelligence and Other Cognitive Functions (eTHINK)
Brief Title: A Study of the Impact of Hemophilia and Its Treatment on Brain Development, Thinking and Behaviour in Children With Hemophilia
Acronym: eTHINK
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-4436; U1111-1202-3415 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-08-21; First posted 2018-09-07 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hemophilia: Children and young adults with hemophilia A or B, all severities, treated in the hemophilia treatment center (comprehensive care) setting, including participation of caregivers/parents completing questionnaires designed to evaluate neurologic, neurocognitive and neurobehavioral function and development.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The participants will undergo a brief physical examination focused on neurologic function (muscle function, sensation, coordination, walking). Parents will be asked by the study team or the psychologist about their children and will complete several commonly used standard surveys about brain development, thinking, behavior, and decision making. The participants will also engage with the psychologist to evaluate development or thinking (IQ), and depending on their age they may be asked to complete one or more commonly used standard surveys about behavior and decision making.

SUMMARY:
The Hemophilia Growth and Development Study (HGDS) nearly 25 years ago showed haemophilia and HIV impacted brain development, thinking, and behaviour in children and adolescents. The eTHINK study is designed to understand whether advances in hemophilia treatment have removed any impact of hemophilia. If there still is an impact of hemophilia, the eTHINK study will help to identify which children or adolescents are still at risk, and how to screen other children. Participants and their child will participate in a comprehensive assessment of child's brain development, thinking and behavior through completing tests and questionnaires. There is only one study visit of 1 to 1.5 hours with no follow-up required

ELIGIBILITY:
Inclusion Criteria: - Male child or young adult (ages 1:0-3:6 and 4:0-21:11 years with diagnosis of congenital hemophilia A or B, any severity, with or without inhibitors - Parent able and willing to provide consent, and young adult with hemophilia (age 18-21) able to provide consent; children (ages 7-14) and adolescents/young adults (ages 14-17) able and willing to provide assent based upon local institutional policies - Parent able and willing to complete neurodevelopment and cognitive parent reported scales during comprehensive or other Hemophilia Treatment Center visit for about 45-60 minutes in English or Spanish depending on age group) - Children, adolescents and young adults with hemophilia (ages 1-21) able to participate in assessments of development and intelligence for about 40-45 minutes and adolescents and young adults (age 11-21) with hemophilia able and willing to complete additional self-assessment scales for about 30-45 minutes during comprehensive or other elective visit for in English or Spanish (depending on age group) - Provision of informed consent before the start of any study-related activities Exclusion Criteria: - Patient aged 3:7-3:11 years (43-47 months) - Prior participation in the study - Prior neurocognitive screening with the same or related instruments in the prior 6 months - Patients with hemophilia or their caregivers for whom test measures may be culturally inappropriate - Patients with hemophilia with known history of alcohol or substance abuse - Patients with hemophilia who have used opiates in the past 24 hours or other illicit drugs within the past 48 hours - Patients with hemophilia currently experiencing an acute bleed that has not resolved - Patients with hemophilia with recent head injury or concussion within the past 4 weeks - Concurrent diagnosis of another bleeding or thrombotic disorder - Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Ages: 1 Year to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults with hemophilia A or B, all severities
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Cognition composite score according to the BAYLEY-III instrument | Day 1
  Normalized score compared to US population (0 = equivalent to US average, negative = below US average, positive = above US average
Behavioural Symptoms Index according to Behavior Assessment System for Children - Third Edition (BASC-3) parent rating scale | Day 1
  Normalized score compared to US population (0 = equivalent to US average, negative = below US average, positive = above US average
Adaptive behaviour domain score according to Adaptive Behavior Assessment System, Third Edition (ABAS-3) rating scale | Day 1
  Normalized score compared to US population (0 = equivalent to US average, negative = below US average, positive = above US average
Global executive composite index according to Behavior Rating Inventory of Executive Function (BRIEF) | Day 1
  Normalized score compared to US population (0 = equivalent to US average, negative = below US average, positive = above US average
Attention and processing speed (full scale IQ) according to Wechsler Preschool and Primary Scale of Intelligence-4th Edition (WPPSI-IV) for age group 4-6 years or Wechsler Abbreviated Scale of Intelligence, 2nd Edition (WASI-II) for age group 7-22 years | Day 1
  Normalized score compared to US population (0 = equivalent to US average, negative = below US average, positive = above US average

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (22):
- United States (22):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Mrakotsky C, Walsh KS, Buranahirun Burns C, Croteau SE, Markert A, Geybels M, Hannemann C, Rajpurkar M, Shapiro KA, Wilkening GN, Ventola P, Cooper DL; eTHINK Study Group. The eTHINK Study: Cognitive and Behavioral Outcomes in Children with Hemophilia. J Pediatr. 2024 Sep;272:114089. doi: 10.1016/j.jpeds.2024.114089. Epub 2024 May 9. PMID 38734133
- [Derived] Buranahirun C, Walsh KS, Mrakotsky C, Croteau SE, Rajpurkar M, Kearney S, Hannemann C, Wilkening GN, Shapiro KA, Cooper DL. Neuropsychological function in children with hemophilia: A review of the Hemophilia Growth and Development Study and introduction of the current eTHINK study. Pediatr Blood Cancer. 2020 Jan;67(1):e28004. doi: 10.1002/pbc.28004. Epub 2019 Oct 8. PMID 31595670